CLINICAL TRIAL: NCT03241810
Title: Randomized Phase 2 Trial of Seribantumab Plus Fulvestrant in Postmenopausal Women With Hormone Receptor-positive, Heregulin Positive (HRG+), HER2 Negative Metastatic Breast Cancer (Merrimack Pharmaceuticals Inc.)
Brief Title: Phase 2 Trial of Seribantumab Plus Fulvestrant in Postmenopausal Women With Metastatic Breast Cancer
Acronym: SHERBOC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Merrimack Inc. terminated the trial early due to business decision
Sponsor: Elevation Oncology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MM-121-02-02-10; 2017-000565-76 (EudraCT Number)
Record Dates: First submitted 2017-08-02; First posted 2017-08-08 (Actual); Results first posted 2020-09-02 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2019-11

CONDITIONS: Metastatic Breast Cancer
Keywords: Breast Cancer, HER2 Negative, Hormone receptor positive
MeSH Terms: conditions — Breast Neoplasms | interventions — seribantumab; Fulvestrant; Histidine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in a 1:1 ratio (experimental arm versus active comparator arm) using an Interactive Web Response System (IWRS). Randomization will be stratified based on bone-only disease (yes, no) and geographic region (US, non-US).
Who Masked: Participant, Care Provider, Investigator
Masking Description: This is a multi-center, randomized, double-blind, placebo-controlled Phase 2 Study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Seribantumab
  Fulvestrant
  Interventions: Drug: Seribantumab; Drug: Fulvestrant
- Arm B (Active Comparator): Placebo
  Fulvestrant
  Interventions: Drug: Fulvestrant; Drug: Placebo

INTERVENTIONS:
Drug: Seribantumab — Seribantumab is a human monoclonal antibody that inhibits ErbB3 signalling
  Other Names: MM-121
  Arms: Arm A
Drug: Fulvestrant — Fulvestrant is an estrogen receptor antagonist with no agonist effects
  Other Names: Faslodex
Drug: Placebo — Placebo
  Other Names: Solution containing 20 mM histidine, 150 mM sodium chloride, at a pH of 6.5
  Arms: Arm B

SUMMARY:
This study is a multi-center, randomized, double-blind, placebo-controlled, Phase 2 study in postmenopausal women with heregulin positive, hormone receptor positive, HER2 negative metastatic, unresectable breast cancer.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled international phase 2 trial in patients with HRG+, HR+, HER2- metastatic breast cancer that has progressed following treatment with no more than 2 prior therapies, one of which must have been a CDK inhibitor. All patients will be screened for heregulin using central testing, and eligible patients will be randomized to receive either seribantumab + fulvestrant or placebo + fulvestrant. Disease status will be assessed according to RECIST v 1.1 to support the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for participation in the study, patients must meet the following criteria. Patients who are HRG negative do not need to complete screening procedures beyond HRG assessment.

1. Patients must have histologically or cytologically confirmed ER+ and/or PR+ (with staining of >1% cells) breast cancer.
2. Patients with confirmed postmenopausal status due to either surgical/natural menopause or ovarian suppression.
3. Patients must be HER2 negative.
4. Patient must have at least one lesion amenable to either core needle biopsy or fine needle aspiration.
5. Patient must have a positive in-situ hybridization (ISH) test for heregulin, as determined by centralized testing of unstained tumor tissue.
6. Patients that have progressed following at least one but no more than two prior systemic therapies in the locally advanced or metastatic disease setting.
7. Patients with documented progression of locally advanced or metastatic disease as defined by RECISTv1.1 (Exception: patients with bone-only metastatic disease are eligible if they have at least 2 lytic lesions visible on a CT or MRI and have documented disease progression on prior therapy based on the appearance of new lesions).
8. Patients with bone-only lesions who have received radiation to those lesions must have documented progression following radiation therapy.
9. ECOG Performance Score (PS) of 0 or 1.
10. Patients with adequate bone marrow reserves.
11. Adequate hepatic function.
12. Adequate renal function.
13. Patient has recovered from clinically significant effects of any prior, surgery, radiosurgery, or other antineoplastic therapy.
14. Patients who have experienced a venous thromboembolic event within 60 days of signing the main consent form should have been treated with anti-coagulants for at least 7 days prior to beginning treatment and for the duration of treatment on this study.

Exclusion Criteria:

Patients must meet all the inclusion criteria listed above and none of the following exclusion criteria.

1. Prior treatment with an anti-ErbB3 antibody.
2. Prior treatment with a chemotherapy in the locally advanced or metastatic disease setting.
3. Patients cannot have received prior treatment with fulvestrant or other SERDs in the locally advanced or metastatic setting.
4. Uncontrolled CNS disease or presence of leptomeningeal disease.
5. Inflammatory breast cancer.
6. History of another active malignancy that required systemic therapy in the last 2 years. Patients with prior history of in-situ cancer, basal, or squamous cell skin cancer are eligible.
7. Patients with an active infection, or unexplained fever > 38.5 C during screening visits or on the first scheduled day of dosing, which in the investigator's opinion might compromise the patients participation in the trial or affect the study outcome. At the discretion of the investigator, patients with tumor fever may be enrolled.
8. Known hypersensitivity to any of the components of seribantumab, fulvestrant, or who have had hypersensitivity reactions to fully human monoclonal antibodies.
9. NYHA Class III or IV congestive heart failure.
10. Patients with a significant history of cardiac disease (i.e. uncontrolled blood pressure, unstable angina, myocardial infarction within 1 year or ventricular arrhythmias requiring medication) are also excluded.
11. Uncontrolled infection requiring IV antibiotics, antivirals, or antifungals; or active human immunodeficiency virus (HIV) infection, active hepatitis B infection or active hepatitis C infection.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Confirmed postmenopausal status due to either surgical/natural menopause or ovarian suppression (initiated at least 28 days prior to Day 1 of Cycle 1).
Enrollment: 22 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Pipas, MD, Study Director — Merrimack Pharmaceuticals Inc.
Locations (59):
- United States (22):
  - Ironwood Cancer and Research Centers- Chandler, Chandler, Arizona
  - Highland Oncology Group, Fayetteville, Arkansas
  - Beverly Hills Cancer Center, Beverly Hills, California
  - Stanford University, Palo Alto, California
  - Saint Helena Hospital, St. Helena, California
  - Stamford Hospital, Stamford, Connecticut
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - UF Health Cancer Center at Orlando Health, Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Columbus Regional Research Institute, Columbus, Georgia
  - Cancer Care Specialists of Central Illinois, Decatur, Illinois
  - James M Stockman Cancer Institute, Frederick, Maryland
  - Holy Cross Hospital Health Center, Silver Spring, Maryland
  - Lahey Clinical Medical Center, Burlington, Massachusetts
  - University of Mississippi, Jackson, Mississippi
  - Mercy Hospital Springfield, Springfield, Missouri
  - Saint Francis Cancer Treatment Center, Grand Island, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Oncology Specialists of Charlotte, Charlotte, North Carolina
  - UPMC Cancer Center, Pittsburgh, Pennsylvania
  - University of Utah Health Care - Huntsman Cancer Institute, Salt Lake City, Utah
- Austria (4):
  - LKH - Universitätsklinikum Graz, Graz
  - Universitaetsklinik fuer Gynaekologie und Geburtshilfe, Innsbruck
  - Krankenhaus der Barmherzigen Schwestern Linz, Linz
  - Medizinische Universität Wien, Vienna
- Belgium (6):
  - Clinique Saint-Pierre, Ottignies, Brabant Wallon
  - Centre Hospitalier de l'Ardenne - Clinique du Sein, Libramont, Luxembourg
  - Universitaire Ziekenhuis Leuven, Leuven, Vlaams Brabant
  - Universitair Ziekenhuis Antwerpen, Antwerp
  - Cliniques Universitaires Saint-Luc, Brussels
  - CHU UCL NAMUR - Sainte Elisabeth, Namur
- Canada (4):
  - University of Calgary, Calgary, Alberta
  - British Columbia Cancer Agency, Kelowna, British Columbia
  - McGill University - Jewish General Hospital, Montreal
  - Centre Hospitalier Affilie Universitaire de Quebec, Québec
- Germany (8):
  - Universitätsklinikum Erlangen, Erlangen, Bavaria
  - Medizinisches Zentrum Bonn Friedensplatz, Bonn
  - Centrum fuer Haematologie und Onkologie Bethanien, Frankfurt
  - Gynäkologisch-Onkologische Praxis Hannover, Hanover
  - Rotkreuzklinikum München-Frauenklinik, Munich
  - Klinikum Rechts der Isar der Technischen Universität München, München
  - Onkologie Rheinsieg, Troisdorf
  - Universitätsklinikum Ulm, Ulm
- Spain (15):
  - Hospital Universitari General de Catalunya, Sant Cugat del Vallès, Barcelona
  - Complejo Hospitalario Universitario La Coruña, A Coruña
  - Hospital Teresa Herrera, A Coruña
  - Hospital Universitari de Girona Doctor Josep Trueta, Girona
  - Complejo Hospitalario de Jaén, Jaén
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Ramón Y Cajal, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Son Llatzer, Palma de Mallorca
  - De La Cruz Merino, Luis, Seville
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At the time of the study termination by the prior Sponsor (Merrimack Pharmaceuticals), 62 sites participated in the study (27 in North America and 35 in Europe).
Groups:
- Arm A (Experimental): Seribantumab and Fulvestrant: Seribantumab (a human monoclonal antibody that targets ErbB3, a cell surface receptor that is activated by the ligand heregulin. Heregulin-driven ErbB3 signaling has been implicated as a mechanism of tumor growth and resistance to targeted, cytotoxic and anti-endocrine therapies. When used in the combination setting, seribantumab is designed to block ErbB3 signaling in order to enhance the anti-tumor effect of a combination therapy partner): fixed dose of 3000 mg intravenously (IV) on day 1 and 15 of each 28-day cycle
  Fulvestrant (a drug treatment of hormone receptor-positive metastatic breast cancer in post-menopausal women with disease progression following anti-estrogen therapy. It is an estrogen receptor antagonist with no agonist effects, which works both by down-regulating and by degrading the estrogen receptor): 500 mg intramuscularly (IM) on Days 1 and 15 of Cycle 1, and then on Day 1 of each subsequent 28 day cycle
- Arm B (Control): Placebo and Fulvestrant: Placebo: intravenously (IV) on day 1 and 15 of each 28-day cycle
  Fulvestrant: (a drug treatment of hormone receptor-positive metastatic breast cancer in post-menopausal women with disease progression following anti-estrogen therapy. It is an estrogen receptor antagonist with no agonist effects, which works both by down-regulating and by degrading the estrogen receptor): 500 mg intramuscularly (IM) on Days 1 and 15 of Cycle 1, and then on Day 1 of each subsequent 28 day cycle
Period: Overall Study
Arm/Group | Arm A (Experimental): Seribantumab and Fulvestrant | Arm B (Control): Placebo and Fulvestrant
Started | 11 | 11
Completed | 11 (Safety population: includes patients receiving at least one dose of study medication.) | 11 (Safety population: includes patients receiving at least one dose of study medication.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients that have signed informed consent, identified as HRG positive based on centralized tissue analysis,& have successfully completed study entry criteria (Safety Population- patients receiving at least one dose of study medication).
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Experimental): Seribantumab and Fulvestrant | Arm B (Control): Placebo and Fulvestrant | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 7 | 15
  >=65 years | 3 | 4 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 11 | 22
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 10 | 9 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: Participants]
  Canada | 0 | 1 | 1
  Belgium | 2 | 1 | 3
  United States | 5 | 6 | 11
  Spain | 4 | 3 | 7
Metastatic burden (TNM Stage at Initial Diagnosis) [Number; unit: Participants] — Based upon the population treated, the most important baseline measure was CT scans to determine metastatic burden, as the primary endpoint was investigator assessed PFS.
  TNM Staging (Tumor size):
  T1 (T1a,T1b & T1c): 2 cm (3/4 of an inch) or less across. T2: > 2 cm but not more than 5 cm (2 inches) across. T3: > 5 cm across. T4 (T4a,T4b,T4c,T4d): Tumor of any size growing into the chest wall or skin. As a rule, the lower the number, the less the cancer has spread. A higher number, such as stage IV, means cancer has spread more. And within a stage, an earlier letter means a lower stage.
  Participants
    TNM Stage I | 0 | 1 | 1
    TNM Stage II | 0 | 2 | 2
    TNM Stage IIa | 4 | 0 | 4
    TNM Stage IIb | 1 | 0 | 1
    TNM Stage III | 0 | 2 | 2
    TNM Stage IIIa | 1 | 0 | 1
    TNM Stage IIIc | 1 | 0 | 1
    TNM Stage IV | 4 | 6 | 10
Heregulin positive status and staining in archival tissue [Count of Participants; unit: Participants] — Women had to be ≥ HRG 1+ positive in their submitted tumor sample to qualify for the study
  Participants | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Progression Free Survival is defined as the time from randomization to the first documented radiographical progression of disease using RECIST v1.1 or death from any cause, whichever comes first as assessed by the investigator.
  The tumor assessment (i.e., scan dates) was used for progression/censor date not the date corresponding to the determination of overall response. Progression-free survival time distribution and median survival for each treatment group were analyzed using the Kaplan-Meier method.
Time Frame: Randomization until progression of disease or death due to any cause up to 13 months (The study terminated prematurely) . The primary analysis was planned to be initiated when 58 PFS events have occurred
Population: Intent-to-Treat (ITT) population treated up to 150 days
Measure: Number; unit: Participants
Arm/Group | Arm A (Experimental): Seribantumab and Fulvestrant | Arm B (Control): Placebo and Fulvestrant
Number analyzed (Participants) | 11 | 11
Participants | 1 | 1

2. Secondary Outcome: Overall Survival
Description: Overall Survival (OS) is defined as the time from the date of randomization to the date of death from any cause. The study was terminated on 30 Nov 2018 . Data represents outcomes up to 150 days of treatment.
Time Frame: Randomization until death due to any cause up to 13 months (The study terminated prematurely)
Population: Intent-to-Treat (ITT) population treated up to 150 days
Measure: Number; unit: participants
Arm/Group | Arm A (Experimental): Seribantumab and Fulvestrant | Arm B (Control): Placebo and Fulvestrant
Number analyzed (Participants) | 11 | 11
participants | 1 | 1

3. Secondary Outcome: Objective Response Rate
Description: Objective Response Rate (ORR) is defined as the proportion of patients with a RECIST v1.1 response recorded from randomization until disease progression characterized as either a Complete Response (CR) or Partial Response (PR) relative to the total number of evaluable patients.
Time Frame: Randomization through end of study up to 13 months (The study terminated prematurely)
Population: Incomplete data for all subjects due to length of time on study treatment and frequency of scanning. All patients analysed had progressive disease. Therefore, they did not meet the criteria for ORR and hence could not be evaluated for CR or PR
Arm/Group | Arm A (Experimental): Seribantumab and Fulvestrant | Arm B (Control): Placebo and Fulvestrant
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Time to Progression
Description: Time to Progression (TTP) is defined as the time from the date of randomization to the date of objective tumor progression.
Time Frame: Randomization to date of objective tumor progression up to 13 months (The study terminated prematurely)
Population: Intent-to-Treat (ITT) population consisted of all participants randomized to the study.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Arm A (Experimental): Seribantumab and Fulvestrant | Arm B (Control): Placebo and Fulvestrant
Number analyzed (Participants) | 11 | 11
days | 52 [33.25 to 72.25] | 48 [34.50 to 58.50]

5. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events Reported With the Combinations of Seribantumab Plus Fulvestrant Versus Fulvestrant Alone
Description: Treatment-emergent adverse events (TEAEs) are defined as any event that occurred after the first dose of study drug and was not present prior to study drug administration or worsened in severity after study drug administration.
Time Frame: TEAEs were collected through the study completion (30 Nov 2018), up to 13 months. Frequency and percent summaries were presented for TEAE defined as adverse events that occur or worsen in severity following the first dose of seribantumab, or fulvestrant
Population: Safety Population: The safety population includes patients receiving at least one dose of study medication. All safety analyses were to be performed on this population.
Measure: Number; unit: participants
Arm/Group | Arm A (Experimental): Seribantumab and Fulvestrant | Arm B (Control): Placebo and Fulvestrant
Number analyzed (Participants) | 11 | 11
participants
  Patients with any TEAE-Related | 7 | 4
  Patients with any TEAE-Serious Adverse event | 1 | 0
  NCI-CTCAE Grade 3 or Higher | 2 | 1

6. Secondary Outcome: Percentage of Treatment-emergent Adverse Events Reported With the Combinations of Seribantumab Plus Fulvestrant Versus Fulvestrant Alone
Description: as for outcome 5
Time Frame: as for outcome 5
Population: Safety Population: The safety population includes patients receiving at least one dose of study medication. All safety analyses were be performed on this population.
Measure: Number; unit: percentage of adverse events
Arm/Group | Arm A (Experimental): Seribantumab and Fulvestrant | Arm B (Control): Placebo and Fulvestrant
Number analyzed (Participants) | 11 | 11
percentage of adverse events
  TEAE-Related | 63.6 | 36.4
  TEAE-Serious Adverse event | 9.1 | 0
  NCI-CTCAE Grade 3 or Higher | 18.2 | 9.1

7. Secondary Outcome: Pharmacokinetic (PK) Profile of Seribantumab When Given in Combination With Fulvestrant and of Fulvestrant When Given in Combination With Serbantumab.
Description: Pharmacokinetic (PK) evaluation are performed on samples obtained pre-dose on day 1 and 15 of each 28-day cycle to assess pre-treatment trough concentrations of MM-121. The maximum observed concentration (Cmax) is presented and calculated usig Non-compartmental analysis (NCA). Serum levels of MM-121 are measured at a central lab using an enzyme-linked immunosorbent assay (ELISA).
Time Frame: The study terminated prematurely after 13 months. Were to be analyzed post-dose on Cycle 1,Week 1 & pre-dose for all subsequent seribantumab infusions until the completion of Cycle 2. Fulvestrant PK samples were to be collected prior to seribantumab dose
Population: Due to the premature study termination, the PK data were not collected. There was no pharmacokinetic data feasible for the analysis, and as such, no related analyses were performed. Hence, data could not be reported in the data table.
Arm/Group | Arm A (Experimental): Seribantumab and Fulvestrant | Arm B (Control): Placebo and Fulvestrant
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From Baseline through to premature study completion up to 13 months (30 Nov 2018)
Description: The safety population includes patients receiving at least one dose of study medication. All safety analyses were be performed on this population. Safety analyses (adverse events and laboratory analyses) were performed using the safety population. Adverse events were coded using the latest MedDRA dictionary (MedDRA 21.0). Severity of adverse events was graded according to the NCI CTCAE version 4.03.
Arm/Group | Arm A (Experimental): Seribantumab and Fulvestrant | Arm B (Control): Placebo and Fulvestrant
All-Cause Mortality (participants affected / at risk) | 10/11 | 10/11
Serious Adverse Events (participants affected / at risk) | 1/11 | 0/11
Other Adverse Events (participants affected / at risk) | 10/11 | 8/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Experimental): Seribantumab and Fulvestrant (N=11) | Arm B (Control): Placebo and Fulvestrant (N=11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Experimental): Seribantumab and Fulvestrant (N=11) | Arm B (Control): Placebo and Fulvestrant (N=11)
Anaemia (Blood and lymphatic system disorders) | 2 | 1
Palpitations (Cardiac disorders) | 1 | 0
Ear Pain (Ear and labyrinth disorders) | 1 | 0
Dry eye (Eye disorders) | 1 | 0
Eye allergy (Eye disorders) | 1 | 0
Lacrimation increased (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 7 | 3
Nausea (Gastrointestinal disorders) | 2 | 3
Dyspepsia (Gastrointestinal disorders) | 3 | 0
Oral pain (Gastrointestinal disorders) | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Stomatitis (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Faeces soft (Gastrointestinal disorders) | 0 | 1
Odynophagia (Gastrointestinal disorders) | 1 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 3 | 1
Fatigue (General disorders) | 2 | 1
Chest discomfort (General disorders) | 0 | 1
Influenza like illness (General disorders) | 1 | 0
Injection site pain (General disorders) | 0 | 1
Injection site reaction (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Hepatomegaly (Hepatobiliary disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Fungal infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperchloraemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 2 | 1
Headache (Nervous system disorders) | 2 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Irritability (Psychiatric disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 1
Urine odour abnormal (Renal and urinary disorders) | 0 | 1
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Hot flush (Vascular disorders) | 2 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Sponsor (Merrimack Pharmaceuticals, INC.) terminated the trial early due to business decision

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-04-28): https://cdn.clinicaltrials.gov/large-docs/10/NCT03241810/Prot_000.pdf
  • Statistical Analysis Plan (2016-01-29): https://cdn.clinicaltrials.gov/large-docs/10/NCT03241810/SAP_001.pdf